CLINICAL TRIAL: NCT04189770
Title: One Plus One Can Be Greater Than Two: Ecological Momentary Assessment for Black Prostate Cancer Survivors and Partners
Brief Title: Lifestyle Behavior Influences Among African American Patients With Stage 0-III Prostate Cancer Survivors and Their Partners
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-0579; NCI-2019-07937 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0579 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cancer Survivor; Partner; Spouse; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, accelerometer, EMA, survey): Patients and partners complete questionnaires over 60 minutes about demographic information, stress, coping, and lifestyle behaviors at baseline and end of study. Patients and partners also receive an accelerometer and complete EMA questionnaire on stress, coping, physical activity, and eating behaviors over 5-10 minutes QID (7:30 am, 11:30 am, 3:30 pm, and 7:30 pm) via an smartphone app for 14 days. Patients and partners also complete a survey on nutrition BIW for a total of 4 surveys.
  Interventions: Device: Accelerometer; Other: Ecological Momentary Assessment; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Device: Accelerometer — Wear accelerometer
Other: Ecological Momentary Assessment — Complete EMA questionnaire
  Other Names: EMA
Other: Questionnaire Administration — Complete questionnaire
Other: Survey Administration — Complete survey

SUMMARY:
This trial studies the day-to-day stress, social support, and health lifestyle behaviors (such as physical activity and nutrition) in African American patients with stage 0-III prostate cancer survivors and their partners. How patients cope with stress may affect their lifestyle behaviors. This study may help understand not only survivors' behaviors but also partners' behaviors and how they interact.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine temporal associations between dyadic coping and health behaviors such as physical activity and diet.

II. Identify social and physical contexts in which health behaviors occur/co-occur among survivors and their partners.

EXPLORATORY OBJECTIVE:

I. Investigate potential moderators for the associations between stress and dyadic coping.

OUTLINE:

Patients and partners complete questionnaires over 60 minutes about demographic information, stress, coping, and lifestyle behaviors at baseline and end of study. Patients and partners also receive an accelerometer and complete Ecological Momentary Assessment (EMA) questionnaire on stress, coping, physical activity, and eating behaviors over 5-10 minutes four time daily (QID; 7:30 am, 11:30 am, 3:30 pm, and 7:30 pm) via an smartphone application (app) for 14 days. Patients and partners also complete a survey on nutrition twice weekly (BIW) for a total of 4 surveys.

ELIGIBILITY:
Inclusion Criteria:

* Survivors are eligible if they self-identify as African American adults
* Had stage 0-III prostate cancer (no restriction on time elapsed since diagnosis)
* Completed adjuvant therapy (i.e., chemo and/or radiation therapy)
* Live together with a current partner/spouse who is eligible for the study
* Do not need physical assistance (e.g., wheelchair, cane)
* Have a smartphone
* Can read and speak English
* Currently are not participating in a health behavior or weight management program
* Men on active surveillance will be included
* Partners are eligible if they are adults
* Partners are eligible if they do not have serious medical conditions (e.g., cancer, congestive heart failure, stroke, and dementia)
* Partners are eligible if they have a smartphone
* Partners are eligible if they can read and speak English
* Partners are eligible if they currently are not participating in a health behavior or weight management program
* The dyad can be either married or unmarried and same-sex or heterosexual

Exclusion Criteria:

* Survivors will be excluded if they had a prior history of other cancer or have metastatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African American prostate cancer survivors and their partners
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Physical activity in both patients and partners | Up to 14 days
  To assess the association between the common dyadic coping of partner or survivor and physical activity of the survivor or partner, will construct 2 new variables corresponding to each common dyadic coping variable for each individual.
Nutrition in both patients and partners | Up to 14 days
  To assess the association between the common dyadic coping of partner or survivor and nutrition of the survivor or partner, will construct 2 new variables corresponding to each common dyadic coping variable for each individual.
Stress in both patients and partners | Up to 14 days
  To assess the association between the common dyadic coping of partner or survivor and nutrition of the survivor or partner, will construct 2 new variables corresponding to each common dyadic coping variable for each individual.
Social and physical contexts where health behaviors occur/co-occur among survivors and partners | Up to 14 days
  Descriptive analysis (e.g., frequency) will be conducted to examine the places (e.g., home, neighborhood) in which the health behaviors occurred and the number of health behaviors engaged alone and with others (especially with partner). Also, contexts (days of a week and times of a day and place) in which survivors and partners engaged in health behaviors together will be investigated. All analyses will be exploratory in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Dalnim Cho, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org